CLINICAL TRIAL: NCT01807182
Title: Cellular Adoptive Immunotherapy Using Autologous Tumor-Infiltrating Lymphocytes Following Lymphodepletion With Cyclophosphamide and Fludarabine for Patients With Metastatic Melanoma
Brief Title: Tumor-Infiltrating Lymphocytes After Combination Chemotherapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sylvia Lee, Associate Professor, Program in Immunology, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2643.00; NCI-2013-00486 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2643.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG9213019 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (TIL, combination chemotherapy, aldesleukin) (Experimental): Patients receive cyclophosphamide IV on days -7 to -6 and fludarabine phosphate IV on days -5 to -1. Patients undergo TIL infusion over 30-60 minutes on day 0 and receive aldesleukin IV every 8 hours on days 1-5 for up to a maximum of 14 doses.
  Interventions: Biological: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Therapeutic Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Therapeutic Tumor Infiltrating Lymphocytes — Undergo TIL infusion
  Other Names: Tumor Infiltrating Lymphocytes

SUMMARY:
This phase II trial studies how well tumor-infiltrating lymphocytes (TIL) after combination chemotherapy works in treating patients with melanoma that has spread to other places in the body. Biological therapies, such as TIL, may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as cyclophosphamide and fludarabine phosphate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving TIL after combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive cyclophosphamide intravenously (IV) on days -7 to -6 and fludarabine phosphate IV on days -5 to -1. Patients undergo TIL infusion over 30-60 minutes on day 0 and receive aldesleukin IV every 8 hours on days 1-5 for up to a maximum of 14 doses.

After completion of study treatment, patients are followed up at 6, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

Step I Inclusion Criteria:

* Stage IV melanoma or stage III melanoma that is unlikely to be cured by surgery
* Able to tolerate high-dose cyclophosphamide, fludarabine and high-dose IL-2
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must have a magnetic resonance imaging (MRI), computed tomography (CT), or positron emission tomography (PET) of the brain within 2 months before consenting if known history of brain metastasis or if clinically indicated; if new lesions are present, principal investigator (PI) or designee should make final determination regarding enrollment
* Patients must have a site of metastatic disease that can be safely resected or biopsied for tissue sufficient for TIL harvest

Step II Inclusion Criteria:

* Patients must have measurable metastatic melanoma
* Able to tolerate high-dose cyclophosphamide, fludarabine, and high-dose IL-2
* ECOG performance status of 0-1
* Patients must have brain imaging by MRI, CT or PET within 30 days prior to lymphodepletion; patients may have asymptomatic brain lesions that are =< 1 cm each, lesions that are > 1 cm that have been irradiated and in the opinion of the investigator no longer represents active disease will also be allowed
* A functional cardiac test (e.g., stress treadmill, stress thallium, multigated acquisition scan (MUGA), dobutamine echocardiogram) to rule out cardiac ischemia within 4 months prior to lymphodepletion is required for all patients
* Pulmonary function tests (PFTs) are required of all patients within 4 months prior to lymphodepletion; forced expiratory volume (FEV)1 and forced vital capacity (FVC) must be >= 65% predicted and diffusion lung capacity for carbon monoxide (DLCO) must be >= 50% predicted
* Patients must have their tumor sent for v-Raf murine sarcoma viral oncogene homolog B1(BRAF) mutational analysis
* Patients must have adequate TIL (at least 40 x 10^6 cells at the pre-expansion stage)

Exclusion Criteria:

Step I Exclusion Criteria:

* Men or women of reproductive ability who are unwilling to use effective contraception or abstinence for 4 months after treatment
* Calculated creatinine clearance (estimated glomerular filtration rate [eGFR]) < 60 ml/min; EGFR values can be determined by either Modification of Diet in Renal Disease (MDRD) or Cockcroft-Gault equation based on the investigator's discretion
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 3 x upper limit of normal
* Total bilirubin > 2.0 mg/dl, except in patients with Gilbert's syndrome whose total bilirubin must not exceed 3.0 mg/dl) deemed by investigator to be irreversible
* FEV1 < 65% predicted, FVC < 65% of predicted, DLCO (corrected for hemoglobin [Hgb]) < 50% predicted); pulmonary function tests (PFTs) within 4 months prior to consent for Step I will be required for patients with underlying risk factors such as smoking history > 10 pack years, or a history of pre-existing symptomatic lung disease (not including melanoma metastases to the lung)
* Pre-existing known cardiovascular abnormalities as defined by any one of the following:

  * Congestive heart failure
  * Clinically significant hypotension
  * Cardiac ischemia, or symptoms of coronary artery disease
  * Presence of cardiac arrhythmias on electrocardiogram (EKG) requiring drug therapy
  * Ejection fraction < 45% (echocardiogram or MUGA), although any patient with an ejection fraction between 45-49% must receive clearance by a cardiologist to be eligible for Step II of the trial
* Clinically significant autoimmune disorders or conditions of immunosuppression; patients with acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV)-1 associated complex or known to be HIV antibody seropositive or known to be recently polymerase chain reaction (PCR)+ for hepatitis B or C are not eligible for this study; the severely depressed or altered immune system found in these patients and the possibility of premature death would compromise study objectives
* Patients with active systemic infection requiring intravenous antibiotics
* Clinically significant psychiatric disease which, in the opinion of the PI or sub-investigator (I), would render immunotherapy and its potential sequelae unsafe or compliance with procedural requirements unlikely

Step II Exclusion Criteria:

* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within 14 days prior to entry; patients of both genders must practice birth control during treatment and for four months after treatment
* Calculated creatinine clearance (eGFR) < 60 ml/min; EGFR values can be determined by either MDRD or Cockcroft-Gault equation based on the investigator's discretion
* AST/ALT > 3 x upper limit of normal
* Total bilirubin > 2.0 mg/dl, except in patients with Gilbert's syndrome whose total bilirubin must not exceed 3.0 mg/dl)
* Clinically significant pulmonary dysfunction (FEV1 < 65% predicted or FVC < 65% of predicted, DLCO (corrected for Hgb) < 50% predicted)
* Pre-existing known cardiovascular abnormalities as defined by any one of the following:

  * Congestive heart failure
  * Clinically significant hypotension
  * Cardiac ischemia, or symptoms of coronary artery disease
  * Presence of cardiac arrhythmias on EKG requiring drug therapy
  * Ejection fraction < 45%, although any patient with an ejection fraction between 45-49% must receive clearance by a cardiologist to be eligible for Step II of this trial
* Absolute neutrophil count less than 1000/mm^3
* Platelet count less than 100,000/mm^3
* Hemoglobin less than 10.0 g/dl
* Untreated central nervous system metastases that are either symptomatic or greater than 1 cm at time of therapy; lesions that are > 1cm that have been irradiated and in the opinion of the PI or sub-I no longer represent active disease may be allowed
* Patients with systemic infections requiring active therapy within 72 hours of lymphodepletion
* Systemic cancer therapy (standard or experimental), including cytotoxic chemotherapy or IL-2, received less than 4 weeks or checkpoint blocking agents (e.g., cytotoxic T-lymphocyte protein [CTLA]-4 or programmed cell death protein [PD]1/PD-ligand [L]1 inhibitors) received less than 6 weeks prior to lymphodepletion, with the exception of targeted therapies
* Commercially available, molecularly targeted therapies (e.g., dabrafenib, trametinib, vemurafenib, imatinib) taken within 7 days prior to lymphodepletion
* Clinically significant autoimmune disorders or conditions of immunosuppression; patients with AIDS or HIV-1 associated complex or known to HIV antibody seropositive or known to be recently PCR+ for hepatitis B or C virus are not eligible for this study; virology testing will be done within 6 months of T cell infusion; the severely depressed or altered immune system found in these patients and the possibility of premature death would compromise study objectives
* Prior treatment with systemic steroids within 4 weeks prior to lymphodepletion (except for physiologic replacement doses for adrenal insufficiency, premedication for contrast allergies for scans, and for drug fever related to targeted therapy)
* Any other significant medical or psychological conditions that would make the patient unsuitable candidate for cell therapy at the discretion of the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia M. Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A patient counts as enrolled on this study when they sign treatment consent on the study. 11 patients signed treatment consent, however 1 patient did not move on to treatment due to increased edema and bleeding at brain metastasis. 10 patients were treated on study.
Groups:
- Treatment (Tumor Infiltrating Lymphocytes (TIL), Combination Chemotherapy, Aldesleukin): Patients receive cyclophosphamide IV on days -7 to -6 and fludarabine phosphate IV on days -5 to -1. Patients undergo TIL infusion over 30-60 minutes on day 0 and receive aldesleukin IV every 8 hours on days 1-5 for up to a maximum of 14 doses.
  Aldesleukin: Given IV
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Therapeutic Tumor Infiltrating Lymphocytes: Undergo TIL infusion
Period: Overall Study
Arm/Group | Treatment (Tumor Infiltrating Lymphocytes (TIL), Combination Chemotherapy, Aldesleukin)
Started | 10
Completed | 7
Not Completed | 3
Not completed — Death | 1
Not completed — New therapy | 1
Not completed — Moved to hospice care | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (TIL, Combination Chemotherapy, Aldesleukin)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Clinical Response Category
Description: Assessed using Response Evaluation Criteria in Solid Tumors 1.1 definitions for complete response, partial response, stable disease, and progressive disease. Clinical response will be determined at 6 weeks, 12 weeks and 24 weeks based on RECIST version 1.137 definitions for Complete Response (CR), Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD). Response reported is best response per participant. A complete response will be defined as total regression of all tumors, a PR as 30% or greater decrease in the sum of the longest diameter of target lesions compared to baseline and PD as 20% increase in the sum of the longest diameter of target lesions compared to the smallest prior diameter (RECIST v1.1 criteria).
Time Frame: Up to 24 weeks post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TIL, Combination Chemotherapy, Aldesleukin)
Number analyzed (Participants) | 10
Participants
  Complete Response | 2
  Partial Response | 2
  Progressive Disease | 2
  Stable Disease | 4

2. Secondary Outcome: Number of Participants Who Experienced in Vivo Persistence of Adoptively Transferred T Cells Following TIL Infusion
Description: Whole exome and RNA sequencing of tumor cells and normal tissue was performed to identify non synonymous missense mutations, which was then used to generate peptide pools to identify neoantigen-reactive T cells. T-Cell Receptor (TCR) sequencing of T cell clonotypes in blood at time of treatment, 10 months and 24 months was performed and used to assess the persistence of a tumor antigen specific clonotype infused in the TIL product.
Time Frame: Up to 24 months
Population: Due to the technical challenges and costs of examining persistence of unmodified TIL cells that do not have a unique tag, the persistence has not been performed in the other patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TIL, Combination Chemotherapy, Aldesleukin)
Number analyzed (Participants) | 1
Participants
  At time of treatment | 1
  10 months post infusion | 1
  24 months post infusion | 1

3. Secondary Outcome: Count of Participants Who Experienced Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Time Frame: Adverse events will be collected through 4 weeks after T cell infusion. Beginning 4 weeks after the T cell infusion, only study-related toxicities will be collected for up to 1 year following T cell infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TIL, Combination Chemotherapy, Aldesleukin)
Number analyzed (Participants) | 10
Participants | 10

4. Secondary Outcome: A Count of Participants With Biomarker Expression Above Threshold
Description: Several biomarkers, CXCL13+ CD4 cells, CXCL13+ CD8+ cells, and regulatory cells were evaluated to assess correlation with clinical responses to TIL therapy.
Time Frame: Up to 24 weeks
Population: Samples from 6 patients were evaluated in depth. Biomarker studies were not performed in all patients due to funding constraints.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TIL, Combination Chemotherapy, Aldesleukin)
Number analyzed (Participants) | 6
Participants
  CXCL13+ as % of CD4 T Cell (40% Threshold) | 2
  Treg as % of CD4 T Cell (40% Threshold) | 3
  CXCL13+ as % of CD8 T Cell (40% Threshold) | 6

ADVERSE EVENTS:
Time Frame: Adverse events will be collected through 4 weeks after T cell infusion. Beginning 4 weeks after the T cell infusion, only study-related toxicities will be collected for up to 1 year following T cell infusion.
Description: All adverse events will be recorded and graded according to the NCI CTCAE version 4.0.
Arm/Group | Treatment (TIL, Combination Chemotherapy, Aldesleukin)
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TIL, Combination Chemotherapy, Aldesleukin) (N=10)
Atrial Fibrulation (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TIL, Combination Chemotherapy, Aldesleukin) (N=10)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 9 (9)
Neutrophil count decreased (Investigations) | 10 (10)
Platelet count decreased (Investigations) | 10 (10)
White blood cell decreased (Investigations) | 9 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 8 (8)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT01807182/Prot_SAP_000.pdf